CLINICAL TRIAL: NCT01442402
Title: Impact of APOL1 Gene Variants in African American Kidney Transplant Recipients: A Study of Clinical Outcomes and Molecular Mechanisms
Brief Title: APOL1 Gene Variants in African American Kidney Transplant Recipients
Status: Terminated | Type: Observational
Why Stopped: Lack of funding/resources
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anil K. Chandraker, MD, Medical Director of Renal Transplantation, Brigham and Women's Hospital
Other Study IDs: 2011P000734
Record Dates: First submitted 2011-09-27; First posted 2011-09-28 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Transplant;Failure,Kidney; Kidney Disease; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Aims 1 and 2:
  Subjects will collect a saliva specimen in an Oragene®•DNA sample collection kit for genotyping. We will also collected any discarded (no longer utilized for clinical purposes) tissue from biopsies.
  Aim 3:
  Prior to transplant, subjects will collect saliva in an Oragene®•DNA sample collection kit for genotyping and 10cc of blood will be drawn into a Na heparin collection tube for APOL1 protein analysis. When applicable, plasmapheresis effluent will be collected. We will also collected any discarded (no longer utilized for clinical purposes)tissue from biopsies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2 APOL1 genotypes: African American transplant recipients with homozygous APOL1 gene variants
- 0 or 1 APOL1 genotypes: African American transplant recipients without homozygous APOL1 gene variants

SUMMARY:
Aim 1:

Determine if there is an association between the APOL1 risk variants and allograft survival and function in African Americans

Aim 2:

Determine if there is an association between the presence of APOL1 risk variants in an African American kidney transplant recipient and the risk of recurrent disease

Aim 3:

Investigate mechanisms of APOL1 associated kidney disease by prospectively following African American kidney transplant recipients throughout their clinical course.

ELIGIBILITY:
Aim 1:

Inclusion Criteria:

* self-reported African American
* 18 years or older
* kidney transplant within 12 years

Aim 2:

Inclusion Criteria for patients with recurrent disease:

* self-reported African American
* 18 years or older
* kidney transplant within 12 years
* recurrent or de novo glomerular disease on allograft kidney biopsy

Inclusion Criteria for control group:

* self-reported African American
* 18 years or older
* kidney transplant within 12 years
* end stage kidney disease due to glomerular nephritis, clinically diagnosed or by native kidney biopsy

Exclusion Criteria for control group:

* clinical evidence of recurrent disease (presence of proteinuria, hematuria, Creatinine >2)

Aim 3:

Inclusion Criteria:

* self-reported African American
* 18 years or older
* scheduled living kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African American Renal Transplant Patients
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Allograft survival | year 1, 3, 5

SECONDARY OUTCOMES:
Allograft function as measured by serum creatinine | creatinine levels at year-1, year-3 and year-5

CONTACTS AND LOCATIONS:
Overall Officials: Anil K Chandraker, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States